CLINICAL TRIAL: NCT06632756
Title: Positive Psychotherapy for Smoking Cessation: A Focus on Strengths to Improve Self-efficacy and Enable Successful Quitting Strategies
Brief Title: Positive Psychology for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Joelle Ferron, Assistant Professor, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2202130-2
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Mental Illness; Tobacco Dependence
MeSH Terms: conditions — Mental Disorders; Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Positive Recovery Smoking Cessation (Individual and Group) (Experimental): The "Positive Recovery for Smoking" program is a 16-week treatment that focuses on the use of identifying signature character strengths and identifying, creating, and enjoying positive life events to facilitate recovery from smoking addiction. The first 4 individual sessions will focus on a self-evaluation of strengths and a focus on the individuals top 5 "signature strengths". The participants will then learn about how their signature strengths currently help them function and when and how they can use these strengths to recover from smoking.
  The group sessions will begin at 5 weeks (following 4 individual sessions) - sessions are structured to begin with a check-in where patients identify their most used signature strengths and take inventory of their smoking and cessation efforts from the past week. We will then support participants in their efforts to learn new ways to navigate positive recovery.
  Interventions: Behavioral: Individual and Group Treatment for Smoking Cessation

INTERVENTIONS:
Behavioral: Individual and Group Treatment for Smoking Cessation — Positive psychology-based individual treatment and groups

SUMMARY:
This study will examine how Positive Psychotherapy (PPT) may help people interested in quitting smoking, quit.

DETAILED DESCRIPTION:
This project aims to adapt the Positive Psychotherapy (PPT) practice for smoking cessation in adults with severe mental illness (SMI), testing its usability, feasibility, and acceptability in a mixed-methods feasibility pilot study. Qualitative interviews will be conducted to obtain usability and acceptability input on the adapted PPT manual from 4-5 Peer Providers. Then, in partnership with The Mental Health Center of Greater Manchester (MHCGM), 6-8 adult smokers with SMI will be recruited who want to quit smoking in the next month and are willing to use nicotine replacement therapy (NRT). The 16-week PPT adaptation ("Positive Recovery for Smoking") will be tested progress on cessation assessed through interviewer-administered quantitative assessments at baseline, 8, and 16 weeks. Self-reported cigarettes per day (CPD) and carbon monoxide (CO) will be collected prior to each group treatment session. Informed by the weekly group check-in of cessation progress (quitting status), qualitative interviews will be conducted at 16 weeks to obtain a more nuanced description of the uptake of the intervention, successful quitting strategies, and barriers to cessation with this new method. The manual and materials will be adapted based on the feedback from the first group and another group of 6-8 participants will be recruited to receive the refined intervention and protocol. The result of this feasibility pilot will provide data on the adapted PPT's feasibility and acceptability, alongside a deep description of strategies used and why and how the treatment was perceived as useful or not to the enrolled participants.

ELIGIBILITY:
Inclusion Criteria:

* age 21+;
* Serious Mental Illness (SMI) diagnosis;
* smoking ≥10 CPD;
* breath CO ≥10;
* desire to quit in the next month;
* willingness to use NRT daily;
* English speaking and literate to engage in the treatment.

Exclusion Criteria:

* legal guardian;
* active substance use disorder.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Abstinence from Smoking | baseline to 16 weeks
  At least 20% of participants will achieve abstinence (0 cigarettes per day and CO less than 6) at 16 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- The Mental Health Center of Greater Manchester, Manchester, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No